CLINICAL TRIAL: NCT04316065
Title: A Randomized, Open-label, Single-dose, 2-sequence, 2-period, Crossover Clinical Trial to Investigate the Bioequivalence Between YHP1906 Tab. 5 mg and YHR1902 Tab. 5 mg in Healthy Volunteers
Brief Title: Bioequivalence Study Between YHP1906 Tab. 5 mg and YHR1902 Tab. 5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Collaborators: Metro Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP1906-101
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): 15 subjects, Cross-over, Single dose of comparator on day 1, Single dose of YHP1906 on day 8
  Interventions: Drug: YHP1906; Drug: YHR1902
- Group 2 (Other): 15 subjects, Cross-over, Single dose of YHP1906 on day 1, Single dose of comparator on day 8
  Interventions: Drug: YHP1906; Drug: YHR1902

INTERVENTIONS:
Drug: YHP1906 — YHP1906 Tab. 5 mg
Drug: YHR1902 — Comparator. YHR1902 Tab. 5 mg

SUMMARY:
A randomized, open-label, single-dose, 2-sequence, 2-period, crossover clinical trial to investigate the bioequivalence between YHP1906 Tab. 5 mg and YHR1902 Tab. 5mg in healthy volunteers

DETAILED DESCRIPTION:
30 healthy subjects will be randomized to one of the 2 groups in the same ratio.

Subjects in group 1 will be administered "comparator" and "YHP1906 Tab. 5 mg" by cross-over design on day 1, 8.

Subjects in group 2 will be administered "YHP1906 Tab. 5 mg" and "comparator" by cross-over design on day 1, 8

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 and above with body mass index(BMI) between 18.5 and 30.0 kg/m2
2. Acceptable medical history, physical examination and laboratory tests during screening
3. Subjects who has signed a written informed consent voluntarily, prior to any procedure, using a form that is approved by the local Institutional Review Board after detailed explanation of the purpose, contents, and characteristic of the drug

Exclusion Criteria:

1. History of clinically significant disease
2. Administration of ETC(ethical-the-counter drug) within 2 weeks or OTC(over-the-counter drug) within 1 week prior to the first dosing
3. Have AST(GOT) and/or ALT(GPT) and/or GGT(γGT) and/or Total Bilirubin > 1.5 times of normal upper limit
4. Volunteers considered not eligible for the clinical trial by the investigator
5. Administration of other investigational products within 6 months prior to the first dosing

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-36 hours
  Area under the plasma drug concentration-time curve [AUCt] of Apixaban
Maximum plasma concentration [Cmax] | 0-36 hours
  Maximum plasma concentration [Cmax] of Apixaban

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-36 hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of Apixaban
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-36 hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] of Apixaban
Time of peak concentration [Tmax] | 0-36 hours
  Time of peak concentration [Tmax] of Apixaban
Terminal phase of half-life [t1/2] | 0-36 hours
  Terminal phase of half-life [t1/2] of Apixaban

CONTACTS AND LOCATIONS:
Overall Officials: Sungdae Kwon, Principal Investigator — Metro Hospital
Locations (1):
- Metro Hospital, Anyang-si, Gyeonggi-do, South Korea